CLINICAL TRIAL: NCT05912322
Title: A Comprehensive in Vivo Evaluation of Aronia Melanocarpa (Michx.) Elliott Bio Juice on Blood Pressure Levels and Endothelial Damage
Brief Title: Evaluation of Black Chokeberry Bio Juice on Blood Pressure Levels and Endothelial Damage
Acronym: AROBLENDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Collaborators: ASCAR Cardiology Clinic, Timisoara City Hospital (Other)
Responsible Party: Principal Investigator, Minodora Andor, MD, PhD, Associate Professor, ASCAR Cardiology Clinic, Timisoara City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5DOC/1425/03.02.2020
Record Dates: First submitted 2022-10-01; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Essential Hypertension; Endothelial Dysfunction; Inflammation
Keywords: black chokeberry; cardiovascular effects; essential arterial hypertension; endothelial dysfunction
MeSH Terms: conditions — Essential Hypertension; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black chokeberry juice (Experimental): 100ml black chokeberry juice/day
  Interventions: Dietary Supplement: Black chokeberry juice
- Control (No Intervention): Lifestyle changes. No juice

INTERVENTIONS:
Dietary Supplement: Black chokeberry juice — 100ml black chokeberry juice/day
  Arms: Black chokeberry juice

SUMMARY:
In Romania, the diseases of the circulatory system account for 59.3% of deaths, representing the main cause of morbidity and mortality.

Barriers of current pharmacological treatments materialized in side effects and limited actions on risk factors increase the necessity of finding more effective, multi-target and less toxic therapeutic strategies. Considering the well-known benefits, natural compounds represent a very important source for drug candidates.

The latest in vitro and in vivo studies on Aronia melanocarpa (Michx.) Elliott have highlighted its antioxidant, anti-inflammatory, anti-proliferative, anti-atherosclerotic, hypotensive, antiplatelet, lipid and glucose reduction properties, making it an excellent candidate for the prevention and treatment of cardiovascular and metabolic disorders.

The aim of this study is to comprehensive evaluate (in vivo) the Aronia melanocarpa bio juice, obtained from Romania on blood pressure levels and endothelial damage.

DETAILED DESCRIPTION:
Patients at risk of developing hypertension (HTN) or suspicion of HTN will be invited for a visit in the Cardiology Clinic of Timisoara City Hospital. After performing the investigations for the suspicion of HTN in the Clinic, the diagnosis of HTN (>140/90mmHg) or pre-HTN (130-139/85-89mmHg) will be made after 24h monitorization, based on the results of Ambulatory Pressure Monitoring Device(ABPM). In function of the results and the patients' risk factors, a treatment strategy (pharmacological or non-pharmacological) will be implemented. Patients who fit the inclusion criteria will be asked to join the study. Study design: Prospective study of 3 months period. The included patients (≈ 100 patients) will be randomized (1:1) in two groups (one receiving 100ml black chokeberry juice (AMJ)/day and one control group, both under lifestyle changes), matched be age, sex and characteristics. The complete list of analysis and investigations will be performed at the inclusion of the study (T0), after 3 months (T3) of non-pharmacological treatment. Periodical phone calls (each 4 weeks) will be made by the clinical pharmacist to assess the health status, adherence, eventual problems of the treatment or difficulty to accomplish the targets. If any of the included patients will develop problems during the proposed treatment (ex: higher blood pressure levels) they will be excluded from the study and classical pharmacological treatment will be applied.

Investigations: familial and personal history of cardiovascular (CV) disease/renal disease and associated risk factors; smoking/drinking/substance abuse/dietary habits, blood pressure measurements, heart rate, weight, height, 12-lead electrocardiography, echocardiography (cardiac, vascular and abdominal), carotid intima-media thickness (IMT), flow mediated vasodilation (FMD), laboratory evaluation of venous blood samples (morning, fasting state >8h harvested on anticoagulant) and urine analysis. The complete blood count, electrolytes, hepatic, renal, lipid, triglycerides and glucose profile of venous blood sample and the urine analysis will be performed by routine laboratory analysis in the Cardiology Clinic. Quantification of several special markers of endothelial injury will be performed, such as: pentraxin-3, soluble endoglin (sEng), endothelin-1; asymmetric dimethylarginine (ADMA). The imagistic investigations will be performed by the same certified cardiologist.

ELIGIBILITY:
Inclusion Criteria:

* informed consent form signed,
* BP values: 130 - 159 / 85 - 99 mmHg (high normal BP and grade 1 HTN) at low-moderate CV risk (a calculated SCORE=1-5%)
* under no concomitant medications

Exclusion Criteria:

* refusal to participate,
* BP ≥ 140/90mmHg with high CV risk,
* acute/chronic administration of any pharmacological treatment during the study period,
* other CV or cerebrovascular pathologies,
* congenital disorders,
* liver/renal diseases,
* history/presence of peptic ulcer,
* acute/chronic inflammatory conditions,
* hypersensibility to black chokeberry juice,
* diabetes mellitus,
* gout,
* pregnancy/breast feeding mother

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Normalization of blood pressure levels | 3 months
  By inhibition of angiotensin I-converting enzyme (ACE). Measurements performed at the same hour/once a day (expressed in mmHg)

SECONDARY OUTCOMES:
Change in systemic and endothelial inflammation | 3 months
  Modification in the values of the special markers that were assessed: pentraxin-3, soluble endoglin (expressed in ng/mL)
Normalization of metabolic profile | 3 months
  glucose, uric acid (expressed in mg/dL)
Normalization of lipid profile | 3 months
  LDL-cholesterol, HDL-cholesterol, total cholesterol, triglycerides (expressed in mg/dL)
Modification in BMI | 3 months
  The weight (expressed in kg) and height (expressed in meters) will be combined to report BMI (body mass index expressed in bk/m^2)
Modification of ADMA | 3 months
  The levels of asymmetric dimethylarginine (ADMA) will be assessed and expressed in mcg/L.

CONTACTS AND LOCATIONS:
Locations (1):
- ASCAR Cardiology Clinic of Timisoara City Hospital, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jurikova T, Mlcek J, Skrovankova S, Sumczynski D, Sochor J, Hlavacova I, Snopek L, Orsavova J. Fruits of Black Chokeberry Aronia melanocarpa in the Prevention of Chronic Diseases. Molecules. 2017 Jun 7;22(6):944. doi: 10.3390/molecules22060944. PMID 28590446
- [Background] Buda V, Andor M, Antal D, Ardelean F, Pavel IZ, dehelean C, Soica C, Folescu R, Andrei F, Danciu C. Cardioprotective effects of cultivated black chokeberries (Aronia spp.): traditional uses, phytochemistry and therapeutic effects. Bioactive Compounds in Nutraceutical and Functional Food for Good Human Health. Ed:IntechOpen 2020, DOI: 10.5772/intechopen.92238, ISBN 978-1-83880-888-4
- See also: European Commission Statistics (2018). Cardiovascular diseases statistics. — http://ec.europa.eu/eurostat/statistics-explained/index.php/Cardiovascular_diseases_statistics#Deaths_from_cardiovascular_diseases